CLINICAL TRIAL: NCT02418806
Title: Group Therapy for Caregivers of Alzheimer's Disease Patients in Spanish Elderly Persons Centres
Acronym: cuiDem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelonabeta Brain Research Center, Pasqual Maragall Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cuiDem/FBB-0113
Record Dates: First submitted 2015-02-06; First posted 2015-04-16 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Family Caregivers; Psychotherapy Group
MeSH Terms: conditions — Alzheimer Disease | interventions — Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Therapy group with follow up sessions (Experimental): Weekly psychotherapy groups during 4 months with a monthly follow up period (12 months)
  Interventions: Behavioral: Psychotherapy groups
- Therapy group without follow up sessions (Experimental): Weekly psychotherapy groups during 4 months
  Interventions: Behavioral: Psychotherapy groups
- Active comparator group (Active Comparator): Weekly self-help groups during 4 months with a monthly follow up period (12 months)
  Interventions: Behavioral: Self-help groups

INTERVENTIONS:
Behavioral: Psychotherapy groups
  Arms: Therapy group with follow up sessions; Therapy group without follow up sessions
Behavioral: Self-help groups
  Arms: Active comparator group

SUMMARY:
An experimental study designed to test the effectiveness of a psychological intervention based on group therapy for the caregivers of Alzheimer's disease patients. The intervention consists of 16 sessions of a cognitive-behavioral psychological group therapy. This study aims to demonstrate that Alzheimer's patients' caregivers can decrease the feelings of burden after been involved in a group therapy.

ELIGIBILITY:
Inclusion Criteria:

* Main caregiver of an Alzheimer Disease Patient.
* Alzheimer Disease Patient with mild/severe cognitive impairment.
* High compliance to therapy sessions.
* Sign informed consent.

Exclusion Criteria:

* Low commitment to develop all study phases.
* Caregiver activity remunerated.
* Caregiver with psychiatric disorders that can affect the development of the sessions.
* Caregivers who have received psychological care during last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of group therapy in caregiver burden measured by Zarit Burden Interview. | 16 months

SECONDARY OUTCOMES:
Change in caregiver burden from baseline compared to the control and active arms measured by Zarit Burden Interview. | 4 months and 16 months
Change in anxiety and depression from baseline compared to the control and active arms measured by Goldberg Scale. | 4 months and 16 months
Descriptive analysis of the caregivers' characteristics (sociodemographics, relation wih the AD patient). | Baseline (0 months)
Descriptive analysis of the caregiver's cognition using DEM-DETECT Module 1. | 4 months
Preliminary cost-effectiveness analysis related resources needed to caregivers and Alzheimer patients. | 4 months - 16 months
Change in quality of life from baseline compared to the control and active arms measured by Casp-19 and SF-36 questionnaires. | 4 months - 16 months
Change in resilience from baseline compared to the control and active arms measured by Connor-Davidson Resilience Scale. | 4 months - 16 months
Change in functional social support from baseline compared to the control and active arms using Duke-UNC questionnaire. | 4 months - 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Poudevida, Psychologist, Principal Investigator — BarcelonaBeta Brain Research Center
Locations (11):
- Spain (11):
  - AFA Barcelona, Barcelona
  - Centro de día Vitalia, Barcelona
  - AFA Burgos, Burgos
  - AFA Castellón, Castellon
  - AGUAFA, Guadassuar
  - AFA Lleida, Lleida
  - Centro de envejecimiento saludable, Málaga
  - Fundació Ana Ribot, Pallejà
  - AVAN, Sabadell
  - AFATE, Santa Cruz de Tenerife
  - AFA Terres de l'Ebre, Tortosa

REFERENCES:
- See also: Pasqual Maragall Foundation website — http://fpmaragall.org/
- See also: BarcelonaBeta Brain Research Center website — http://www.barcelonabeta.org/